CLINICAL TRIAL: NCT03490123
Title: Defining the Best Distribution Strategy of Azithromycin for Yaws Eradication (The Yaws 3 Trial)
Brief Title: Evaluation of an Intensive 3-round MDA Strategy Towards Yaws Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lihir Medical Centre (Other)
Collaborators: Barcelona Institute for Global Health (Other); National Department of Health of Papua New Guinea (Unknown); World Health Organization (Other); University of Masarykova (Unknown); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Oriol Mitja, MD, PhD, Lihir Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yaws3
Record Dates: First submitted 2018-03-29; First posted 2018-04-06 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Yaws
Keywords: Azithromycin; Endemic treponematoses; Mass drug administration; Eradication; Papua New Guinea
MeSH Terms: conditions — Yaws | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Community intervention study
Who Masked: Outcomes Assessor
Masking Description: Data collection teams separate from the teams responsible for MDA and screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Repeated total community treatment, TCT with study drug: Azithromycin tablets, 30mg/Kg (maximum 2g), a single dose every 6 months, for 12 months (3 doses).
  Study interventions are:
  R1-Total community treatment with azithromycin, R2-Total community treatment with azithromycin, R3-Total community treatment with azithromycin.
  Interventions: Drug: R1-Total community treatment with azithromycin; Drug: R2-Total community treatment with azithromycin; Drug: R3-Total community treatment with azithromycin
- Control (Active Comparator): Single total community treatment, TCT, with study drug: Azithromycin tablets, 30mg/Kg (maximum 2g), a single, at month 0 (1 dose); followed by two total targeted treatment, TTT, with study drug: Azithromycin tablets, 30mg/Kg (maximum 2g), a single, at months 6 and 12.
  Study interventions are:
  R1-Total community treatment with azithromycin, R2-Total targeted treatment with azithromycin, R3-Total targeted treatment with azithromycin.
  Interventions: Drug: R1-Total community treatment with azithromycin; Drug: R2-Total targeted treatment with azithromycin; Drug: R3-Total targeted treatment with azithromycin

INTERVENTIONS:
Drug: R1-Total community treatment with azithromycin — At month 0, all study participants (regardless of their yaws status) will receive 30 mg/Kg (maximum 2 g) of azithromycin orally under direct observation. Benzathine benzylpenicillin will be reserved as a backup for patients who cannot be treated with AZI, and who are not allergic to penicillin.
  Other Names: R1-TCT
Drug: R2-Total community treatment with azithromycin — At month 6, all study participants (regardless of their yaws status) will receive 30 mg/Kg (maximum 2 g) of azithromycin orally under direct observation. Benzathine benzylpenicillin will be reserved as a backup for patients who cannot be treated with AZI, and who are not allergic to penicillin.
  Other Names: R2-TCT
  Arms: Intervention
Drug: R3-Total community treatment with azithromycin — At month 12, all study participants (regardless of their yaws status) will receive 30 mg/Kg (maximum 2 g) of azithromycin orally under direct observation. Benzathine benzylpenicillin will be reserved as a backup for patients who cannot be treated with AZI, and who are not allergic to penicillin.
  Other Names: R3-TCT
  Arms: Intervention
Drug: R2-Total targeted treatment with azithromycin — At 6 months, study participants will be screened for active yaws. Participants with yaws and their contacts will receive 30 mg/Kg (maximum 2 g) of azithromycin orally under direct observation. Benzathine benzylpenicillin will be reserved as a backup for patients who cannot be treated with AZI, and who are not allergic to penicillin.
  Other Names: R2-TTT
  Arms: Control
Drug: R3-Total targeted treatment with azithromycin — At 12 months, study participants will be screened for active yaws. Participants with yaws and their contacts will receive 30 mg/Kg (maximum 2 g) of azithromycin orally under direct observation. Benzathine benzylpenicillin will be reserved as a backup for patients who cannot be treated with AZI, and who are not allergic to penicillin.
  Other Names: R3-TTT
  Arms: Control

SUMMARY:
The current principle of yaws eradication (the Morges strategy) is based on single round mass drug administration (MDA) of azithromycin (AZI) called total community treatment (TCT) followed by targeted treatment of active cases every 6 months to detect and treat cases and contacts called total targeted treatment (TTT). Studies done in Papua New Guinea (PNG) show that 1 round of MDA will probably not suffice to stop transmission of infection. It may be preferable to conduct 3 rounds of MDA prior to the switch to TTT because of high coverage requirements to achieve elimination, particularly of latent cases. The investigators plan to determine whether 3 rounds of MDA are more effective for reaching yaws elimination. This research is needed to guide national programmatic implementation and needs to be done as soon as possible to scale up the program in the country.

The aim of this proposal is to ascertain the number of rounds of MDA with AZI to be included in an improved strategy towards yaws eradication. The study will be implemented in 38 wards of New Ireland Province (NIP). The investigators will compare two different distribution strategies of MDA: (A) strategy with 3 biannual rounds of MDA and (B) a single mass treatment round of MDA followed by targeted treatment of cases and contacts. The investigators will also monitor the risk of appearance of antimicrobial resistance in Treponema pertenue.

DETAILED DESCRIPTION:
In 2013 WHO piloted the yaws eradication MDA strategy in several countries, including PNG. A study carried out on Lihir Island has shown that 1-round MDA with single-dose oral AZI reduced the prevalence of yaws by 90% at 12-months. However, this did not suffice to stop transmission of infection. At baseline, the estimated prevalence of PCR-confirmed active infection was 1.8% and greatly reduced to 0.4% at 6-months, and 0.1% at 24 months; but prevalence increased again to 0.4% at 42 months after MDA. The relapse of untreated latent infections appeared to hinder elimination efforts in this community. Almost half of subjects with newly identified active yaws cases during follow up targeted treatment programs reported having not been present for MDA. T. p. pertenue may become resistant to macrolide antibiotics, as has occurred with T. p. pallidum (the causative agent of syphilis) in some developed countries, which necessitates close monitoring for the emergence of resistance. The investigators recently reported the first documented genotypic macrolide resistance in T. p. pertenue infections in PNG. A total of five clinical specimens, out of 208 samples tested during the post-MDA period of 3·5 years, demonstrated a T. p. pertenue strain carrying the A2059G point mutation. There was only local spread of the resistant clone among relatives and friends and further spread was immediately stopped through the use of alternative (benzathine penicillin) antibiotic to treat the newly identified cases and contacts.

The eligible population will be people targeted for MDA treatment living in the three LLG study areas at time of implementation. The 38 wards will be randomly assigned (1:1) to receive 1 vs 3 rounds of MDA using AZI. All villages within a ward will receive the same intervention in an effort to minimize contamination between villages. The intervention arm will receive 3 rounds (0, 6, 12 months) of MDA with AZI, each round known as total community treatment (TCT); control arm will receive 1 round (0 months) of MDA with AZI followed by total targeted treatment (TTT) (6 and 12 months). During each MDA round all study participants will receive 30 mg/Kg (maximum 2 g) of AZI orally under direct observation.

The primary outcome will be prevalence of PCR-confirmed active yaws measured in the entire population at 18 months. The investigators will estimate the evolution of latent yaws prevalence measured as the proportion of children 1-15 years who are dually positive on the DPP test at two time-points (0, 18 months).

ELIGIBILITY:
Inclusion Criteria:

* all people resident or not in wards in the study region present at time of implementation or in subsequent surveys

Exclusion Criteria:

* Children younger than 6 months
* Known allergy to macrolide antibiotics
* Refusal at village or individual levels

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56000 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of active and of latent yaws at 18 months | 18 months
  Prevalence of active yaws confirmed by PCR at 18 months and prevalence of latent yaws determined by reaginic and non-reaginic positive DPP tests at 18 months

SECONDARY OUTCOMES:
Appearance of macrolide resistant yaws strains across the study population | 18 months
  T. p. pertenue molecular analyses

CONTACTS AND LOCATIONS:
Locations (1):
- Namatanai Rural Hospital, Kavieng, New Ireland Province, Papua New Guinea

IPD SHARING:
Plan to Share IPD: Undecided
Possible statistical and modelling exercises

REFERENCES:
- [Background] Mitja O, Godornes C, Houinei W, Kapa A, Paru R, Abel H, Gonzalez-Beiras C, Bieb SV, Wangi J, Barry AE, Sanz S, Bassat Q, Lukehart SA. Re-emergence of yaws after single mass azithromycin treatment followed by targeted treatment: a longitudinal study. Lancet. 2018 Apr 21;391(10130):1599-1607. doi: 10.1016/S0140-6736(18)30204-6. Epub 2018 Feb 7. PMID 29428183
- [Background] Mitja O, Houinei W, Moses P, Kapa A, Paru R, Hays R, Lukehart S, Godornes C, Bieb SV, Grice T, Siba P, Mabey D, Sanz S, Alonso PL, Asiedu K, Bassat Q. Mass treatment with single-dose azithromycin for yaws. N Engl J Med. 2015 Feb 19;372(8):703-10. doi: 10.1056/NEJMoa1408586. PMID 25693010
- [Derived] John LN, Beiras CG, Houinei W, Medappa M, Sabok M, Kolmau R, Jonathan E, Maika E, Wangi JK, Pospisilova P, Smajs D, Ouchi D, Galvan-Femenia I, Beale MA, Giacani L, Clotet B, Mooring EQ, Marks M, Vall-Mayans M, Mitja O. Trial of Three Rounds of Mass Azithromycin Administration for Yaws Eradication. N Engl J Med. 2022 Jan 6;386(1):47-56. doi: 10.1056/NEJMoa2109449. PMID 34986286